CLINICAL TRIAL: NCT01824199
Title: CYP2C19 Genotype as a Predictor of Gastric Acid Suppression and Healing of Erosive Esophagitis
Brief Title: CYP2C19 Genotype Predictor of Gastric Acid Suppression
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Katzka, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-008053
Record Dates: First submitted 2013-03-27; First posted 2013-04-04 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Esophagitis
Keywords: Esophagitis
MeSH Terms: conditions — Esophagitis | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omeprazole (Experimental): Patients will undergo whole blood testing for CYP2C19 genotype and will be started on omeprazole 40 mg once daily in the morning 30 minutes before breakfast. The Mayo Dysphasia Questionnaire 30 day (MDQ-30day) will be used during the study. At the end of 8 weeks, patients will undergo dual probe pH/impedance testing on therapy and a clinically indicated endoscopy to rule out Barrett's esophagus and assess healing. CYP2C19 genotyping will be performed in the Mayo laboratory.
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Omeprazole — Patients with LA Grade B-D erosive esophagitis identified at the time of endoscopy will be prospectively recruited. Patients will undergo whole blood testing for CYP2C19 genotype and will be started on omeprazole 40 mg once daily in the morning 30 minutes before breakfast. The Mayo Dysphasia Questionnaire -30 day (MDQ-30day) will be used during the study. At the end of 8 weeks, patients will undergo dual probe pH/impedance testing on therapy and a clinically indicated endoscopy to rule out Barrett's esophagus and assess healing. CYP2C19 genotyping will be performed in the Mayo laboratory.
  Other Names: Prilosec

SUMMARY:
If CYP2C19 genotype can predict the efficacy of healing erosive esophagitis and gastric acid secretion in patients taking once a day omeprazole.

DETAILED DESCRIPTION:
Proton pump inhibitors are metabolized through the CYP2C19 hepatic enzyme system. Several variant genotypes of this enzyme exist which may lead to decreased, normal or increased metabolism of the proton pump inhibitor. With alteration of metabolism, the degree of gastric acid suppression achieved and efficacy in treating reflux could be affected. For example, Asian populations who have low activity of CYP2C19, commonly need lower doses of proton pump inhibitors to manage gastroesophageal reflux because of more sustained blood levels and availability of the drug. Theoretically, those patients who are rapid metabolizers would receive less effective treatment with proton pump inhibitors

ELIGIBILITY:
Inclusion criteria:

* Age 18 or older
* Have either mild-to-moderate Los Angeles (LA) Classification System grade B, moderately severe LA grade C, or severe LA grade D erosive reflux esophagitis
* Or patients having a clinically indicated pH/impedance monitoring on proton pump inhibitor therapy for indications of gastroesophageal reflux disease.

Exclusion criteria:

* Neoplasm of the esophagus or stomach
* Use of drugs that interfere with CYP2C19 metabolism Diazepam, phenytoin, amitriptyline, clomipramine, clopidogrel Cyclophosphamide, progesterone, fluoxetine, fluvoxamine, ketoconazole Lansoprazole, omeprazole, ticlopidine
* Evidence of active H. pylori infection
* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy
* Disorders which predispose to unreliable responses such as Schizophrenia, Alzheimer's disease or significant memory loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03 (Estimated); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The correlation specific to CYP2C19 genotype with gastric acid suppression by omeprazole. | 8 weeks

SECONDARY OUTCOMES:
To assess patients gastrointestinal symptoms, in patients with EoE by means of standard validated questionnaires | 30 days
  trouble swallowing, heartburn, acid regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: David Katzka, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States